CLINICAL TRIAL: NCT02855801
Title: Exercise Training in Patients With Rheumatoid Arthritis and Cryotherapy: Feasibility Study
Brief Title: Exercise Training in Patients With Rheumatoid Arthritis and Cryotherapy
Acronym: RhumatEx
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P/2012/139
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-08

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Cryotherapy; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- constant exercise without cryotherapy (Experimental): constant exercise without cryotherapy
  Interventions: Other: constant exercise
- constant exercise with cryotherapy (Experimental): constant exercise with cryotherapy
  Interventions: Other: constant exercise; Other: cryotherapy
- intermittent exercise, no cryotherapy (Experimental): intermittent exercise without cryotherapy
  Interventions: Other: intermittent exercise
- intermittent exercise and cryotherapy (Experimental): intermittent exercise with cryotherapy
  Interventions: Other: cryotherapy; Other: intermittent exercise

INTERVENTIONS:
Other: constant exercise
  Arms: constant exercise with cryotherapy; constant exercise without cryotherapy
Other: cryotherapy
  Arms: constant exercise with cryotherapy; intermittent exercise and cryotherapy
Other: intermittent exercise
  Arms: intermittent exercise and cryotherapy; intermittent exercise, no cryotherapy

SUMMARY:
The main objective of this project is to study, in patients with rheumatoid arthritis, the effects of an intermittent type exercise associated with cryotherapy on the level of inflammation during its recovery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >18 years old, < 80 years old
* Signature of informed consent for participation
* Affiliation to a social security scheme or French beneficiary of such a regime.
* confirmed rheumatoid arthritis and monitoring by the rheumatology department of the University Hospital of Besancon.
* If there is a corticosteroid therapy, it must be stable for at least 1 month and less than or equal to 10 mg of prednisone equivalent per day
* Clinical and biological activity will be moderate (ie not in remission and not severe based on Disease Activity Score 28 joints - DAS 28 - to be between 2 and 6
* Patients could be treated with DMARDs (Disease-Modifying Drugs).

Exclusion Criteria:

* Patient under guardianship, curatorship, under judicial protection, major incapable
* Patients whose body mass index (BMI) greater than 30,
* Pathology incompatible with the completion of a cycle ergometer exercise (heart, vascular, respiratory, orthopedic ...)
* Change in DAS28 greater than 1.2 in the previous 3 months Inclusion
* A patient with a DAS28 > 6
* about the cold: Raynaud's syndrome, cold known allergy, sickle cell anemia, cryoglobulinemia, uncontrolled hypertension
* Patient unable to follow protocol because of cognitive, psychiatric or language difficulties.
* Inability to follow protocol for causes related to health problems (unrelated Rheumatoid Arthritis) or socio-professional.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
plasma concentration of C-reactive protein | 48 hours after the end of the exercise

CONTACTS AND LOCATIONS:
Overall Officials: Clement Pati, MD, Principal Investigator — CHRU Besancon
Locations (1):
- Centre Hospitalier Régional Universitaire, Besançon, Franche-Comté, France

IPD SHARING:
Plan to Share IPD: No